CLINICAL TRIAL: NCT06460766
Title: Validity and Reliability of the Inflammatory Arthritis Facilitators and Barriers to Physical Activity (IFAB) Questionnaire for Individuals With Pediatric Rheumatic Disease
Brief Title: Validity and Reliability of the Inflammatory Arthritis Facilitators and Barriers to Physical Activity Questionnaire
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nilay Arman, Assistant Professor, Istanbul University - Cerrahpasa
Other Study IDs: Z651y2FQ
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Rheumatic Diseases; Pediatric ALL; Children, Only
Keywords: pediatric rheumatic disease; physical activity; juvenile idiopathic arthritis; juvenile dermatomyositis; juvenile fibromyalgia syndrome
MeSH Terms: conditions — Rheumatic Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Motor Activity; Arthritis, Juvenile; Dermatomyositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
No tool has been found to evaluate behaviors that may hinder or facilitate physical activity in individuals with pediatric rheumatic diseases. In this sense, the importance of examining physical activity barriers and facilitators in children with rheumatic diseases is clear. We believe that our study will guide the increase in physical activity, which is very important for reducing disease risks in individuals with pediatric rheumatic diseases. The aim of our study is to examine the validity and reliability of the Inflammatory Arthritis Facilitators and Barriers to Physical Activity (IFAB) Questionnaire in individuals with pediatric rheumatic diseases (juvenile idiopathic arthritis, juvenile fibromyalgia syndrome, juvenile dermatomyositis).

DETAILED DESCRIPTION:
Children and adolescents with rheumatic diseases can experience significant disability in both the short and long term due to pain, muscle weakness, fatigue, and restricted joint movement. Exercise training has been noted to potentially benefit individuals with pediatric rheumatic diseases by alleviating various clinical symptoms related to physical disability. In this regard, it is important to routinely assess and monitor physical inactivity and sedentary behaviors, along with examining behaviors that may hinder or facilitate physical activity. However, no tool has been encountered to assess behaviors that may hinder or facilitate physical activity in individuals with pediatric rheumatic disease. In this sense, the importance of examining physical activity barriers and facilitators in children with rheumatic disease is clear. The Inflammatory Arthritis Facilitators and Barriers to Physical Activity (IFAB) questionnaire was developed to assess perceived facilitators and barriers to physical activity in patients with inflammatory arthritis. For this purpose, the validity and reliability of the IFAB questionnaire in individuals with pediatric rheumatic diseases (juvenile idiopathic arthritis, juvenile fibromyalgia syndrome, juvenile dermatomyositis) will be examined. Under the supervision of a physical therapist, participants will be assessed using the IFAB questionnaire to evaluate perceived facilitators and barriers to physical activity, the Fear Avoidance Beliefs Questionnaire - Physical Activity (FABQ-PA) questionnaire for fear-avoidance beliefs, and the Motivation Scale For Participation In Physical Activity (MSPPA) to measure motivation for physical activity participation. The results of the IFAB questionnaire will be utilized in the validity and reliability analysis, as well as in the analysis of construct validity. For reliability analysis, the IFAB questionnaire will be repeated after 7 days. All forms will be sent to children in Google form format. It is planned to include 70 children in this study. Factor analysis methods will be used in the analysis of the factor structure of the scale, correlation analyses (Pearson and Spearman coefficients) will be used in the analysis of validity and test-retest reliability. Cronbach's alpha analysis will be used in the reliability analysis. The study will be the first to examine physical activity barriers and facilitators in Turkish children with rheumatic disease. The results will contribute to the identification of physical activity barriers and facilitators in Turkish children with rheumatic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer
* 12-18 ages
* Diagnosed with juvenile idiopathic arthritis, juvenile dermatomyositis and juvenile fibromyalgia syndrome by a pediatric rheumatologist
* Residing in Turkey

Exclusion Criteria:

* Having a vision or hearing problem
* Difficulty adhering to the treatment program

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric rheumatic patients aged 12-18 years who meet the inclusion criteria will be included in our study.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Inflammatory Arthritis Facilitators and Barriers to Physical Activity (IFAB) Questionnaire (Time Frame: Change from baseline to 7 day) | Time Frame: Change from baseline to 7 day
  To assess the perceived facilitators and barriers of physical activity in patients with inflammatory arthritis, the IFAB Questionnaire, developed by Davergne et al. The IFAB consists of 10 items measuring factors that either encourage or hinder physical activity. The total score ranges from 70 to 70, a high score indicates a higher level of facilitators and/or a lower level of barriers. In our study, patient's perceived facilitators and barriers to physical activity will be evaluated with IFAB.
Fear Avoidance Beliefs Questionnaire-Physical Activity (FABQ-PA) | Baseline
  The fear-avoidance beliefs related to physical activity and work effects in low back pain were developed by Waddell et al. The physical activity section consists of 5 questions, with the first question not included in scoring. Each question is evaluated on a scale of 0-6, and patients can score a minimum of 0 and a maximum of 24 points. In our study, patient's fear avoidance beliefs will be evaluated with FABQ-PA.
Motivation Scale For Participation In Physical Activity (MSPPA) | Baseline
  MSPPA was developed by Tekkursun Demir and Cicioglu. It was developed to assess children's motivation to participate in physical activity. The scale, which consists of 16 items, is in the 5-point Likert type. In our study, patient's motivations about physical activity will be evaluated with MSPPA.

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Arman, Asst. Prof., Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No